CLINICAL TRIAL: NCT06916026
Title: A Comparison of Immediate Implant Placement With Deproteinized Bovine Bone vs Deproteinized Bovine Bone With HAM Gel as Space Filling Material: A Randomized Controlled Trial.
Brief Title: Immediate Implant Placement With Deproteinized Bovine Bone vs Deproteinized Bovine Bone With HAM Gel
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: immediate implant placement
Record Dates: First submitted 2025-02-14; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-01

CONDITIONS: Badly Broken Down Vital Teeth
Keywords: Immediate implant placement; jumping gap; xenograft; Bone healing; Human amniotic membrane; bovine bone graft
MeSH Terms: interventions — Transplantation, Heterologous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: blinding of outcome assessors and participants will be achieved as the different outcomes will be assessed for all groups by assessors other than the researchers doing the procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Xenograft (Active Comparator): Gap distance grafting using xenograft.
  Interventions: Procedure: Xenograft
- Xenograft mixed with HAM gel. (Active Comparator): Gap distance grafting using xenograft mixed with HAM gel.
  Interventions: Procedure: Xenograft mixed with HAM gel.

INTERVENTIONS:
Procedure: Xenograft — Gap distance grafting using xenograft
  Arms: Xenograft
Procedure: Xenograft mixed with HAM gel. — Gap distance grafting using xenograft mixed with HAM gel.
  Arms: Xenograft mixed with HAM gel.

SUMMARY:
Statement of the problem: Immediate implant placement is faced with several problems. One of the most important is the jumping gap present after implant placement and whether it needs to be augmented or not.

Aim: The aim of this study is to compare the effect of xenograft to xenograft mixed with HAM gel for grafting of the jumping gap in immediate implant placement in the molar region.

DETAILED DESCRIPTION:
Aim: The aim of this study is to compare the effect of xenograft to xenograft mixed with HAM gel for grafting of the jumping gap in immediate implant placement in the molar region.

Materials and Methods: This parallel arm, randomized controlled clinical trial will involve systemically free patients with remaining roots or badly decayed teeth in the posterior region requiring implant placement. They will be randomly allocated to two equal groups. Group A (control group, n=12) will receive immediate implants (grafting with xenograft), and group B (test group, n=12) will receive immediate implants (grafting with xenograft& HAM). After implant placement, buccal bone thickness (1ry outcome), bone density (2nd outcome) and implant stability will be assessed (2nd outcome). The parameters will be assessed at baseline, 6 and 12 months. Postoperative pain and swelling will be recorded daily by the patient for the 1st two weeks post surgically. Postoperative medication will be prescribed to the patient and postoperative instructions will be explained in detail. Follow-up will be performed to assess the parameters and to ensure performing proper oral hygiene. Data collected will be tabulated and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old, with non-restorable first and second molars indicated for immediate implant placement in both arches.
* Patient who are medically free patients (American Society of Anesthesiologists I; ASA I)
* Minimum remaining alveolar height of four to six millimeters distance from the apex of the socket to the floor of maxillary sinus for maxillary teeth and minimum remaining alveolar height of six millimeters distance from the apex of the socket to the inferior alveolar nerve for mandibular teeth.
* Minimum alveolar Bucco-palatal dimension of 7 mm.

Exclusion Criteria:

* Patients with known systemic diseases which can affect normal bone formation or blood coagulation.
* Patients who are smokers.
* Presence of signs of active infection or pus formation.
* Absence or loss of buccal wall prior to implant placement.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Buccal bone thickness | At Baseline , Six months & 12 months
  assessment of the buccal bone thickness using cone beam computed tomography (CBCT) in mm

SECONDARY OUTCOMES:
Implant stability | at baseline,6 and 12 months
  using Ostell

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of oral and dental medicine , Suez university, Suez, Suez Governorate, Egypt